CLINICAL TRIAL: NCT03430089
Title: Safety of a Single Dose (Participants Aged 9 Years and Older) or Two Doses Given 28 Days Apart (Participants Aged 6 Months to 8 Years) of the Shenzhen Quadrivalent Influenza Vaccine (Split Virion), Inactivated
Brief Title: Safety of a Single Dose or Two Doses of Shenzhen Quadrivalent Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FSQ01; U1111-1174-4615 (Other: WHO Universal Trial Number)
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Influenza; Flu
Keywords: Influenza; Flu
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Phase I-like, open-label, descriptive, monocenter study, which includes 5 groups of participants of varying ages and doses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1: 6 to 35 months (Experimental): Shz QIV 0.25 mL, 2 doses
  Interventions: Biological: Shz QIV 0.25 mL, 2 doses
- Group 2: 3 to 8 years (Experimental): Shz QIV 0.5 mL, 2 doses
  Interventions: Biological: Shz QIV 0.5 mL, 2 doses
- Group 3: 9 to 17 years (Experimental): Shz QIV 0.5 mL, single dose
  Interventions: Biological: Shz QIV 0.5 mL, single dose
- Group 4: 18 to 60 years (Experimental): Shz QIV 0.5 mL, single dose
  Interventions: Biological: Shz QIV 0.5 mL, single dose
- Group 5: 61 years and older (Experimental): Shz QIV 0.5 mL, single dose
  Interventions: Biological: Shz QIV 0.5 mL, single dose

INTERVENTIONS:
Biological: Shz QIV 0.25 mL, 2 doses — Administered intramuscularly in the anterolateral aspect of the thigh in infants (aged 6 to 12 months) or into the deltoid muscle (participants aged more than 12 months), 28 days apart.
  Arms: Group 1: 6 to 35 months
Biological: Shz QIV 0.5 mL, 2 doses — Administered intramuscularly into the deltoid muscle, 28 days apart
  Arms: Group 2: 3 to 8 years
Biological: Shz QIV 0.5 mL, single dose — Administered intramuscularly into the deltoid muscle.
  Arms: Group 3: 9 to 17 years; Group 4: 18 to 60 years; Group 5: 61 years and older

SUMMARY:
This phase I-like, open-label, monocenter, descriptive, single-arm clinical safety study will investigate the Shenzhen quadrivalent influenza vaccine (Shz QIV) in 100 participants aged 6 months and older in China.

Participants aged 9 years or more will receive a single dose of Shz QIV, and participants aged 6 months to 8 years will receive two doses of Shz QIV administered 28 days apart.

DETAILED DESCRIPTION:
Healthy participants will either receive a single dose (participants 9 years or older) or two doses (participants 6 months to 8 years) of the Shz QIV. Safety in terms of serious adverse events, solicited injection site and systemic reactions, and unsolicited adverse events will be collected before and 28 days after each and any dose.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 6 months on the day of inclusion
* For participants aged 6 months through 17 years: Informed consent form has been signed and dated by the parent(s) or another legally acceptable representative, if applicable. Additionally an assent form has been signed and dated by the participant if aged 8 through 17 years (based on local regulations) For participants aged 18 years and older: Informed consent form has been signed and dated by the participant
* Participant / Participant and parent/legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures
* For participants aged less than 2 years only: Born at full term of pregnancy (≥37 weeks) and with a birth weight ≥ 2.5 kg

Exclusion Criteria:

* Participant is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile
* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination [or the first trial vaccination]) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine or planned receipt of any vaccine within the period from 4 weeks before study vaccination (or the first study vaccination) to 4 weeks following study vaccination (or the last study vaccination)
* Previous vaccination against influenza with either the study vaccine or another vaccine from the current season
* Receipt of any vaccine or planned receipt of any vaccine within the period from 2 weeks before trial vaccination (or the first trial vaccination) to 2 weeks following trial vaccination (or the last trial vaccination)
* For participants aged 6 to 8 years only: Previous vaccination against influenza vaccine in the past
* For participants aged 9 years and older: Previous vaccination against influenza (in the previous 6 months) with either the trial vaccine or another vaccine
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Self-reported thrombocytopenia or known thrombocytopenia as reported by the parent/legally acceptable representative, contraindicating IM vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (axillary temperature ≥ 37.1°C). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of serious adverse reactions or Grade 3 non-serious adverse reactions following vaccination with Shz QIV | Within 28 days after vaccination
  Number of participants reporting serious adverse reactions and Grade 3 adverse reactions following a vaccination with Shz QIV

SECONDARY OUTCOMES:
Occurrence of unsolicited systemic AEs reported in the 30 minutes following vaccination/each and any vaccination | Within 30 minutes after vaccination
Occurrence of solicited (prelisted in the subject diary and the electronic Case Report Form [CRF]) injection site reactions and systemic reactions occurring between D0 and D7 after vaccination/each and any vaccination | Up to 7 days after vaccination
Occurrence of unsolicited (spontaneously reported) AEs from D0 to D28 after vaccination/each and any vaccination | Up to 7 days after vaccination
Occurrence of SAEs | Up to 56 days after the 1st vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Investigational Site 002, Xishuangbanna Dai Autonomous Prefecture, Yunnan, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Liu X, Park J, Xia S, Liang B, Yang S, Wang Y, Syrkina O, Lavis N, Liu S, Zhao C, Ding J, Hu J, Samson SI, de Bruijn IA; FSQ01 and FSQ02 Study Groups. Immunological non-inferiority and safety of a quadrivalent inactivated influenza vaccine versus two trivalent inactivated influenza vaccines in China: Results from two studies. Hum Vaccin Immunother. 2022 Nov 30;18(6):2132798. doi: 10.1080/21645515.2022.2132798. Epub 2022 Nov 3. PMID 36328438
- See also: Related info — http://www.sanofipasteur.com